CLINICAL TRIAL: NCT04969159
Title: Insulin Resistance in Septic Patients in the Acute Phase and After Discharge From Hospital
Brief Title: The Degree, Duration and Frequency of Insulin Resistance in Non-operated Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Jens Rikardt Andersen (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, Primary Investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: insulin - sepsis
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Sepsis
Keywords: septicaemia; insulin resitance; continous blood glucose
MeSH Terms: conditions — Sepsis; Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — standard treatment in the clinical routine

SUMMARY:
Surgery induces insulin resistance lasting for 2-3 weeks. We wanted to elucidate if stress-metabolic, medical conditions carry the same effect.

DETAILED DESCRIPTION:
Background: Insulin resistance is well documented after surgery in a severity positively correlated to the degree of trauma (Thorell et al. 1999; Chambrier et al. 2000). Similar phenomena have been described in severely ill patients in ICU with consequences for the survival (Van den Berghe et al. 2001; The NICE-SUGAR Study Investigators 2009). The documentation, however, is scarce and the extent is unknown in acutely ill patients with sepsis.

Method: Adult, consecutive, non-diabetic patients with elevated CRP, leukocyte counts, SOFA-score of ≥ 2 were monitored with fasting p-C-peptide, blood glucose, CRP, leukocyte count and HOMA-IR at admittance, discharge and at two follow-up visits 2 weeks and 4 weeks after admission. Blood glucose levels were measured continuously during the whole study period with a flash glucose monitor mounted on the patients' upper arm. The diagnosis was sepsis, urosepsis, pneumonia, erysipecosis, bacteremia, infection with unknow focus and covid-19.

ELIGIBILITY:
Inclusion Criteria:

* elevated CRP on acute asdmission
* elevated leukocyte count on admission
* SOFA-score ≥ 2
* diagnosis: bacterial sepsis
* full age and authority

Exclusion Criteria:

* not able to understand the protocol
* not able to co-operate
* diabetes mellitus of any kind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adults acutely admnitted to hospital with diagnosed sepsis on bacterial basis or on basis of covid-19
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
continous blood glucose | 4 weeks
  flash glucose monitor on the upper arm

SECONDARY OUTCOMES:
C-peptide | 4 weeks
  plasma concentration
HOMA-IR | 4 weeks
  calculated glucose load test

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, MD,MPA, Study Director — University of Copenhagen
Locations (1):
- Department of endocrinology, Slagelse Hospiatl, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: No
no plans